CLINICAL TRIAL: NCT00527137
Title: An Open-label, Randomized, Non-inferiority Study of Novel Erythropoiesis Stimulating Protein (NESP) and Recombinant Human Erythropoietin (rHuEPO) for the Treatment of Anemia in Pediatric Subjects With Chronic Renal Insufficiency (CRI) or End-stage Renal Disease (ESRD) Receiving Dialysis
Brief Title: NESP Pediatric Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20000100
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Pre-dialysis; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Darbepoetin alfa

ARMS (2):
- rHuEPO (Active Comparator)
  Interventions: Drug: rHuEPO
- darbepoetin alfa (Experimental)
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa — Dose 100U rHuEPO = 0.42 mcg NESP; adjust as necessary (+/- 25% of the starting dose) to maintain Hb withing 10.0 - 12.5 g/dL
  Arms: darbepoetin alfa
Drug: rHuEPO — same as previous rHuEPO dose at randomization; adjust as necessary (+/- 25% of the starting dose) to maintain Hb withing 10.0 - 12.5 g/dL
  Arms: rHuEPO

SUMMARY:
Open-label, randomized study of NESP in pediatric subjects 18 years of age or younger. Subjects will receive study drug (NESP or rHuEPO) for 28 weeks after a 2 week screening and baseline period. During the study, procedures include bloodwork for laboratory assessments and vital signs. Dose titration determined by hemoglobin values taken weekly during the study. Antibody samples taken at baseline and during the end of study assessments. A physical examination and laboratory tests will conclude the study.

ELIGIBILITY:
Inclusion Criteria:

* 1 to 18 years of age
* ESRD receiving dialysis or CRI with eGFR less than 30 mL/min
* Baseline hemoglobin 9.5 - 12.5 g/dL and iron replete
* Stable rHuEPO therapy for 8 weeks

Exclusion Criteria:

* Scheduled for a living-related kidney transplant
* Uncontrolled blood pressure
* seizure activity
* Hyperparathyroidism
* Major surgery within 12 weeks or active inflammatory disease
* Currently receiving antibiotics
* Clinical evidence of malignancy
* Pregnant or breast-feeding

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2000-08; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
To demonstrate that NESP is comparable (not inferior) to rHuEPO for the treatment of anemia in pediatric subjects with CRI or ESRD receiving dialysis | Entire Study

SECONDARY OUTCOMES:
To determine the safety and tolerability of NESP in the treatment of anemia in the pediatric population with CRI or ESRD | Entire Study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Warady BA, Arar MY, Lerner G, Nakanishi AM, Stehman-Breen C. Darbepoetin alfa for the treatment of anemia in pediatric patients with chronic kidney disease. Pediatr Nephrol. 2006 Aug;21(8):1144-52. doi: 10.1007/s00467-006-0071-0. Epub 2006 May 25. PMID 16724235
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com